CLINICAL TRIAL: NCT03527095
Title: A Phase 1, Open-label, Randomised, Cross Over Study to Compare the Pharmacokinetics of Different Oral Formulations of FDL169 in Healthy Subjects Following Single Doses
Brief Title: A Study to Compare the Pharmacokinetics of Different Oral Formulations of FDL169 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Flatley Discovery Lab LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FDL169-2017-06
Record Dates: First submitted 2018-05-04; First posted 2018-05-16 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Regimen A (Experimental): FDL169 200 mg reference tablet
  Interventions: Drug: FDL169
- Regimen B (Experimental): FDL169 200 mg testing tablet 1
  Interventions: Drug: FDL169
- Regimen C (Experimental): FDL169 200 mg testing tablet 2
  Interventions: Drug: FDL169
- Regimen D (Experimental): FDL169 200 mg testing tablet 1 or 2 with high fat diet
  Interventions: Drug: FDL169
- Regimen E (Experimental): FDL169 200 mg testing tablet 1 or 2, fasted
  Interventions: Drug: FDL169
- Regimen F (Experimental): FDL169 200 mg testing tablet 1 or 2, with standard diet
  Interventions: Drug: FDL169

INTERVENTIONS:
Drug: FDL169 — CFTR corrector

SUMMARY:
This is a randomised, cross-over study comprised of 6 periods in healthy subjects.Subjects will receive Regimens A, B and C in a randomised crossover manner in the fed state, followed by Regimens D, E and F in a randomised crossover manner, in the fasted or fed state, as applicable.

DETAILED DESCRIPTION:
This is a single centre, randomised, cross-over study comprised of 6 periods in healthy males and females.Subjects will receive Regimens A, B and C in a randomised crossover manner in the fed state, followed by Regimens D, E and F in a randomised crossover manner, in the fasted or fed state, as applicable.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and non-pregnant, non-lactating female subjects
* Aged 18 to 55 years
* Body mass index of 18.0 to 32.0 kg/m2
* Must agree to the use of an adequate method of contraception

Exclusion Criteria:

* Subjects who have received any IMP in a clinical research study within the previous 3 months
* History of any drug or alcohol abuse in the past 2 years
* Current smokers and those who have smoked within the last 12 months.
* Alkaline phosphatase, aspartate aminotransferase and/or alanine aminotransferase level >1.5 x upper limit of normal at screening
* Abnormal renal function at screening
* Clinically significant abnormal biochemistry, haematology, coagulation profile or urinalysis
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
* History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or GI disease, neurological or psychiatric disorder.
* Subjects with a history of gall stones or abdominal surgery eg cholecystectomy
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
* Subjects who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedy (including known inhibitors or inducers of CYP3A4

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2018-06-21 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability of FDL169 and its metabolites with different formulations | 17 weeks
  To determine the relative bioavailability of FDL169 and its metabolites M1 and M3, following different tablet formulations compared to a reference tablet

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 17 weeks
  Safety and tolerability of FDL169 and its metabolites M1 and M3 , as determined by the incidence of adverse events (Aes) and serious adverse events (SAE)s.
Pharmacokinetic parameters, Cmax | 17 weeks
  The pharmacokinetic parameters of FDL169 and its metabolites M1 and M3 , maximal plasma concentration (Cmax)
Pharmacokinetic parameters, Tmax | 17 weeks
  The pharmacokinetic parameters of FDL169 and its metabolites M1 and M3; maximal concentration (Tmax)
Pharmacokinetic parameters, AUC | 17 weeks
  The pharmacokinetic parameters of FDL169 and its metabolites M1 and M3; area under the plasma concentration curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Ordonez, Study Chair — Flatley Discovery Lab
Locations (1):
- Quotient Sciences, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided